CLINICAL TRIAL: NCT03576313
Title: Mass Drug Administration of Ivermectin and Dihydroartemisinin-piperaquine as an Additional Intervention for Malaria Elimination
Acronym: MASSIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other); National Malaria Control Programme, The Gambia (Other Government); Liverpool School of Tropical Medicine (Other); Radboud University Medical Center (Other); University of Durham (Other); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SCC 1593
Record Dates: First submitted 2018-05-31; First posted 2018-07-03 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Malaria
Keywords: transmission; reduction
MeSH Terms: conditions — Malaria | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: This cluster-randomized trial will involve 32 villages in the Upper River Region of The Gambia that will be randomized to MDA with IVM and DP or to standard of care in a ratio 1:1
Who Masked: Outcomes Assessor
Masking Description: Malaria prevalence will be determined by technicians blinded to the treatment arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention: IVM and DP (Experimental): Mass Drug Administration with ivermectin (IVM) and dihydroartemisinin-piperaquine (DP) will be given to participants in the intervention villages plus the NMCP standard malaria control intervention
  Interventions: Drug: dihydroartemisinin-piperaquine (DP); Drug: ivermectin (IVM); Other: standard malaria control interventions only
- control: standard malaria control intervetions (Active Comparator): Participants in the control clusters will receive only standard malaria control interventions such as Artemether Lumefantrine, LLINs, IRS, SMC and IPTp as implemented by the National Malaria Control Program (NMCP) of the Gambia
  Interventions: Other: standard malaria control interventions only

INTERVENTIONS:
Drug: dihydroartemisinin-piperaquine (DP) — DP will be available as tablets of 320/40mg and 160/20mg piperaquine/ dihydroartemisinin per tablet. Administration of a full course of DP will be done as per manufacturer's guidelines once daily for 3 days and according to body weight. DP will be taken orally with water and without food
  Arms: intervention: IVM and DP
Drug: ivermectin (IVM) — IVM will be available as tablets of 3mg or 6mg strength. It will be given at 300-400μg/kg/day over 3 days (to the nearest whole tablet). IVM will also be taken on an empty stomach with water
  Arms: intervention: IVM and DP
Other: standard malaria control interventions only — this is the standard malaria control interventions in the Gambia

SUMMARY:
This is a community-based cluster-randomized trial in which a novel approach to interrupt residual malaria transmission by mass drug administration (MDA) with ivermectin (IVM) combined with dihydroartemisinin-piperaquine (DP) will be tested. This cluster-randomized trial will involve 32 villages in the Upper River Region of The Gambia that will be randomized to MDA with IVM and DP or to standard of care in a ratio 1:1. This trial aims at establishing whether MDA with IVM and DP can reduce or interrupt malaria transmission in medium to low transmission settings by reducing vector survival and the human reservoir of infection. MDA with IVM and DP will be implemented in the intervention villages and all human settlements in the buffer zone, with the aim of minimizing spillover effects. Control clusters will receive standard malaria control interventions as implemented by the National Malaria Control Program. The primary outcomes will be the prevalence of malaria infection determined by molecular methods in all age groups at the peak of the second transmission season (November-December 2019) and the vector's parous rate 7-14 days after MDA.

DETAILED DESCRIPTION:
The hypothesis of this project is that mass drug administration (MDA) with ivermectin (IVM) and dihydroartemisinin-piperaquine (DP) can reduce or interrupt malaria transmission in medium to low transmission settings by reducing vector survival and the human reservoir of infection. The research questions include the following:

1. Will MDA with IVM plus DP (3 rounds per transmission season) in communities with high coverage of vector control interventions further reduce malaria transmission (up to local elimination)?
2. Will MDA with IVM suppress the vector population?
3. What is the most socially acceptable and sustainable way of achieving and maintaining high coverage of MDA with IVM and DP, and of embedding it within local communities and stakeholders?
4. What is the impact of MDA with IVM on prevalence of ectoparasites and helminths
5. What is the cost and cost-effectiveness of this intervention compared to standard malaria control measures?

ELIGIBILITY:
Inclusion Criteria

* Age/anthropometry

  1. For IVM: weight ≥ 15kg or height ≥90 cm;
  2. For DP: age > 6 months
* Willingness to comply with trial procedures
* Individual written informed consent obtained at the beginning of the study

Exclusion Criteria:

* Exclusion criteria for both IVM and DP will include the following:
* Known chronic illness (eg HIV, TB, hepatitis and severe malnutrition).

Additionally for IVM:

1. Pregnancy (any trimester) and breast feeding
2. Hypersensitivity to IVM
3. Travel to Loa loa endemic countries (e.g. Central Africa)

Additionally for DP:

1. First trimester pregnancy
2. Hypersensitivity to DP
3. Taking drugs that influence cardiac function or prolong QTc interval

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4939 (Actual)
Dates: Start 2018-08-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
prevalence of malaria infection | at 12 months
  Prevalence of malaria infection determined by molecular methods number of participants with a positive varATS quantitative PCR divided by the total number of participants sampled
Vector's parous rate | 7-14 days after mass drug administration (MDA)
  Malaria prevalence will be used as an indicator of on-going malaria transmission, while vector's parous rate will quantify the effect of IVM on vector survival and mosquito population age structure. Proportion: number of parous vectors divided by the total number of collected vectors

SECONDARY OUTCOMES:
malaria prevalence | at 6 months
  malaria prevalence at the peak of the first transmission season of number of participants with a positive varATS quantitative PCR divided by the total number of participants sampled
incidence of clinical (laboratory confirmed) malaria cases | after MDA over 6 months period
  incidence of clinical (laboratory confirmed) malaria cases at health facilities of Number of clinical malaria cases observed divided by person-years of follow-up
serological markers of recent malaria | after MDA over 6 months period
  serological markers of recent malaria infection by Mean Fluorescent Intensity of the different antigens will be determined and presented as a geometric mean
serological markers of recent Anopheles exposure | after MDA over 6 months period
  serological markers of recent Anopheles exposure by Mean Fluorescent Intensity of the different antigens will be determined and presented as a geometric mean
mosquito density | over 24 months after MDA
  Total number of mosquitoes collected during the study period across both intervention and control villages
mosquito mortality | 21 days post treatment
  mosquito mortality after feeding on IVM treated individuals Number of mosquitoes that die after a blood meal 21 days post-treatment divided by total number of mosquitoes blood fed
sporozoite rates in field-caught mosquitoes | over 24 months after MDA
  Number of P. falciparum circumsporozoite antibody (CSP) positive mosquitoes divided by the total number of mosquitoes caught

OTHER OUTCOMES:
drug resistance markers | after MDA 6 months
  prevalence of drug resistance markers in the number of malaria parasites with drug-resistance markers divided by the total number of samples tested

CONTACTS AND LOCATIONS:
Overall Officials: Umberto D'alessandro, MD, PhD, Principal Investigator — MRC @ LSHTM
Locations (1):
- Basse Villages, Basse Santa Su, The Gambia

REFERENCES:
- [Derived] Kositz C, Vasileva H, Mohammed N, Achan J, Dabira ED, D'Alessandro U, Bradley J, Marks M. Risk factors for non-participation in ivermectin and dihydroartemisinin-piperaquine mass drug administration for malaria control in the MASSIV trial. Malar J. 2024 Feb 22;23(1):54. doi: 10.1186/s12936-024-04878-2. PMID 38383367
- [Derived] Fehr A, Nieto-Sanchez C, Muela J, Manneh E, Baldeh D, Ceesay O, D'Alessandro U, Dabira E, Kingori P, Peeters Grietens K, Bardaji A, Bunders-Aelen J, Zuiderent-Jerak T. Doing 'reciprocity work': The role of fieldworkers in a mass drug administration trial in the Gambia. Glob Public Health. 2022 Dec;17(12):4116-4128. doi: 10.1080/17441692.2022.2125998. Epub 2022 Oct 2. PMID 36183416
- [Derived] Dabira ED, Soumare HM, Conteh B, Ceesay F, Ndiath MO, Bradley J, Mohammed N, Kandeh B, Smit MR, Slater H, Peeters Grietens K, Broekhuizen H, Bousema T, Drakeley C, Lindsay SW, Achan J, D'Alessandro U. Mass drug administration of ivermectin and dihydroartemisinin-piperaquine against malaria in settings with high coverage of standard control interventions: a cluster-randomised controlled trial in The Gambia. Lancet Infect Dis. 2022 Apr;22(4):519-528. doi: 10.1016/S1473-3099(21)00557-0. Epub 2021 Dec 15. PMID 34919831
- [Derived] Dabira ED, Soumare HM, Lindsay SW, Conteh B, Ceesay F, Bradley J, Kositz C, Broekhuizen H, Kandeh B, Fehr AE, Nieto-Sanchez C, Ribera JM, Peeters Grietens K, Smit MR, Drakeley C, Bousema T, Achan J, D'Alessandro U. Mass Drug Administration With High-Dose Ivermectin and Dihydroartemisinin-Piperaquine for Malaria Elimination in an Area of Low Transmission With High Coverage of Malaria Control Interventions: Protocol for the MASSIV Cluster Randomized Clinical Trial. JMIR Res Protoc. 2020 Nov 19;9(11):e20904. doi: 10.2196/20904. PMID 33211022